CLINICAL TRIAL: NCT02972385
Title: Pharmacogenomics of Warfarin in Hispanics and Latinos
Status: Recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Jason H Karnes, Assistant Professor, University of Arizona
Other Study IDs: 1608762767
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Thrombosis; Hemorrhage
Keywords: warfarin; blood clotting
MeSH Terms: conditions — Thrombosis; Hemorrhage | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retention: Samples with DNA Description: Isolated DNA will be stored in freezers at minus 80 degrees.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Mouthwash sample — A one time mouthwash sample will be performed.
Procedure: Blood Draw — Patients who are receiving a blood draw during their regular clinical appointment will be asked for a blood sample of 15 milliliters. Genomic DNA will be isolated for genotyping and patient plasma samples will also be stored.

SUMMARY:
Warfarin is a commonly used blood thinner to treat and prevent blood clots. It is important to take the right dose of warfarin because too much can increase the risk of bleeding and too little can increase the risk of blood clots. This is why patients are closely monitored especially when they begin warfarin therapy. When clinicians prescribe warfarin, they have to consider different factors such as patient's age, body size, diet, and other medications that can interact with warfarin.

Certain genes have also been found to affect warfarin dose. Individuals have variations in these genes, which can help explain why some patients need higher dose and others require less. These factors have been used to better predict a patient's warfarin dose requirement. However, these predictions were created based on Caucasian populations and they may not be accurate in predicting a safe warfarin dose if a patient is not Caucasian. This study aims to identify new genetic variation that affects warfarin dosing in Hispanic and Latino populations and try to better predict a Hispanic or Latino patient's warfarin dose requirement.

DETAILED DESCRIPTION:
If the patient is willing to hear about the study, during routine clinical care, one of the patient's providers will approach patients meeting the study criteria about participation in the study. Study personnel will not approach potential participants unless permission is given to the patient's provider. If the patient would like to participate in the study, study personnel will discuss details of the study in person during the patient's routine clinical care visit. There will also be a flyers available for posting and for distribution to potential participants.

Participants consenting to the study will be asked to provide a cheek swab or mouthwash sample to provide buccal cells for DNA extraction. If the patient is receiving a blood draw during their regular clinical appointment, participants will be asked for a blood sample of 15 milliliters. Genomic DNA will be isolated for genotyping and patient plasma samples will also be stored.

Linear regression will be used to test association of SNPs with therapeutic warfarin dose using the algorithms derived by the International Warfarin Pharmacogenomics Consortium. The primary phenotype (weekly stable warfarin dose) will be transformed by square root. SNPs and other variables associated with warfarin dose will be assessed in univariate analyses and entered into stepwise linear regression to determine the adjusted association with dose requirements using R2. Quality control procedures will include deviation from Hardy-Weinberg Equilibrium, and SNP and sample exclusions based on call rates. Ancestry-informative marker (AIM) analysis will be performed to estimate ancestry in each individual.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Ability to give informed consent
* Therapeutic INR for at least 2 consecutive clinic visits
* Self-identifies as Hispanic or Latino

Exclusion Criteria:

* Less than 18 years old
* Unable to give informed consent
* Severe hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be Hispanic and Latino patients on stable doses of warfarin therapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Stable warfarin dose | At time of enrollment
  Dose of warfarin required to maintain stable INR for at least 2 consecutive clinic visits.

CONTACTS AND LOCATIONS:
Locations (1):
- Banner University Medical Center - Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No